CLINICAL TRIAL: NCT04329650
Title: Phase 2, Randomized, Open-label Study to Compare Efficacy and Safety of Siltuximab vs. Corticosteroids in Hospitalized Patients With COVID19 Pneumonia
Brief Title: Efficacy and Safety of Siltuximab vs. Corticosteroids in Hospitalized Patients With COVID-19 Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Judit Pich Martínez (Other)
Responsible Party: Sponsor-Investigator, Judit Pich Martínez, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SILCOR-COVID-19
Record Dates: First submitted 2020-03-31; First posted 2020-04-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — siltuximab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Siltuximab 11mg/Kg (Experimental)
  Interventions: Drug: Siltuximab
- Dexamethasone 6mg/24h (Active Comparator)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Siltuximab — A single-dose of 11mg/Kg of siltuximab will be administered by intravenous infusion.
  Arms: Siltuximab 11mg/Kg
Drug: Dexamethasone — A dose of 6mg/24 hours of dexamethasone during 10 days will be administered orally or by intravenous infusion.
  Arms: Dexamethasone 6mg/24h

SUMMARY:
In our center up to 25% of the hospitalized patients with COVID-19 progress and need an intensive care unit. It is urgent to find measures that can avoid this progression to severe stages of the disease. We hypothesize that the use of anti-inflammatory drugs used at the time they start hyperinflammation episodes could improve symptoms and prognosis of patients and prevent their progression sufficiently to avoid their need for be admitted to an Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Hospitalized patient (or documentation of a hospitalization plan if the patient is in an emergency department) with illness of more than 5 days of duration with evidence of pneumonia by chest radiography / tomography computed chest and meets at least one of the following requirements:

   1. Non-critical patient with pneumonia in radiological progression and / or
   2. Patient with progressive respiratory failure
3. Laboratory confirmed SARS-CoV-2 infection (by PCR) or other commercialized analysis or public health in any sample collected 4 days before the randomization or COVID-19 criteria following the defined diagnostic criteria at that time in the center.
4. Be willing and able to comply with the study related procedures / evaluations.
5. Women of childbearing potential * should have a negative serum pregnancy test before enrollment in the study and must commit to using methods highly effective contraceptives (intrauterine device, bilateral tubal occlusion, vasectomized couple and sexual abstinence).
6. Written informed consent. In case of inability of the patient to sign the informed consent, a verbal informed consent from the legal representative or family witness (or failing this, an impartial witness outside the investigator team) will be obtained by phone.

When circumstances so allow, participants should sign the consent form. The confirmation of the verbal informed consent will be documented in a document as evidence that verbal consent has been obtained.

Exclusion Criteria:

1. Patient who, in the investigator's opinion, is unlikely to survive> 48 hours after the inclusion in the study.
2. Presence of any of the following abnormal analytical values at the time of the inclusion in the study:

   * absolute neutrophil count less than 2000 / mm3;
   * AST or ALT> 5 times the upper limit of normality;
   * platelets <50,000 per mm3.
3. Patients with respiratory support greater than or equal to 60%
4. In active treatment with immunosuppressants or previous prolonged treatment (more 3 months) of oral corticosteroids for a disease not related to COVID-19 at a dose greater than 10 mg of prednisone or equivalent per day.
5. Known active tuberculosis or known history of tuberculosis uncompleted treatment.
6. Patients with active systemic bacterial and / or fungal infections.
7. Patients who have received previous treatment with IL6 inhibitor (tocilizumab, sarilumab).
8. Participants who, at the investigator's discretion, are not eligible to participate, regardless of the reason, including medical or clinical conditions, or participants potentially at risk of not following study procedures.
9. Patients who do not have entry criteria in the Intensive Care Unit.
10. Pregnancy or lactation.
11. Known hypersensitivity to siltuximab or to any of its excipients (histidine, histidine hydrochloride, polysorbate 80 and sucrose).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Proportion of patients requiring ICU admission at any time within the study period. | 29 days

SECONDARY OUTCOMES:
Days of stay in the ICU during the study period. | 29 days
Days until resolution of fever defined as body temperature (axillary ≤ 36.6 ° C, oral ≤ 37.2 ° C, or rectal or tympanic ≤ 37.8 ° C) for at least 48 hours, without administration of antipyretics or until hospital discharge. | 29 days
Proportion of patients with a worsening requirement of supplemental oxygen at 29 days. days. | 29 days
Days with hypoxemia (SpO2 <93% in ambient air or requiring oxygen supplemental or mechanical ventilation support) at 29 days. | 29 days
Proportion of patients using mechanical ventilation at 29 days. | 29 days
Days with use of mechanical ventilation at 29 days. | 29 days
Days until the start of use of mechanical ventilation, non-invasive ventilation or use of high flow nasal cannula (if the patient have not previously required these interventions at the inclusion of the study) at 29 days. | 29 days
Days of hospitalization among survivors at 29 days. | 29 days
Mortality rate from any cause at 29 days. | 29 days
Proportion of patients with serious adverse events at 29 days. | 29 days
Proportion of patients with invasive bacterial or fungal infections clinically significant or opportunistic with grade 4 neutropenia (count neutrophil absolute <500 / mm3) at 29 days. | 29 days
Proportion of patients with invasive bacterial or fungal infections clinically significant or opportunistic at 29 days. | 29 days
Proportion of patients with grade 2 or higher adverse reactions related to the infusion of the sudy treatments at 29 days. | 29 days
Proportion of patients with hypersensitivity reactions of grade 2 or higher related to the administration of the study treatments at 29 days. | 29 days
Proportion of patients with gastrointestinal perforation at 29 days. | 29 days
Proportion of patients with secondary severe infections confirmed by laboratory or worsening of existing infections at 29 days. | 29 days
Changes from baseline in plasma leukocyte levels at days 1, 3, 5, 7 and 9. | Days 1, 3, 5, 7 and 9
Changes from baseline in plasma hemoglobin levels at days 1, 3, 5, 7 and 9. | Days 1, 3, 5, 7 and 9
Changes from baseline in plasma platelet at days 1, 3, 5, 7 and 9. | Days 1, 3, 5, 7 and 9
Changes from baseline in plasma creatinine levels at days 1, 3, 5, 7 and 9. | Days 1, 3, 5, 7 and 9
Changes from baseline in plasma total bilirubin levels at days 1, 3, 5, 7 and 9. | Days 1, 3, 5, 7 and 9
Proportion of patients with ALT≥ 3 times ULN (for patients with initial values normal) or> 3 times ULN AND at least 2 times more than the initial value (for patients with abnormal initial values) at days 1, 3, 5, 7 and 9. | Days 1, 3, 5, 7 and 9
Changes from baseline in plasma biomarkers (PCR, lymphocytes, ferritin, d-dimer and LDH) at days 1, 3, 5, 7 and 9. | Days 1, 3, 5, 7 and 9
Changes from baseline in chest Rx at days 1, 3 and 5. | Days 1, 3 and 5
Analysis of genetic variants in CYP enzymes and transporters SLCO1B1, ABCCs and ABCB1 to the response to the study treatments. | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Felipe García, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (4):
- Spain (4):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitari Mútua de Terrassa, Terrassa

IPD SHARING:
Plan to Share IPD: No